CLINICAL TRIAL: NCT00521547
Title: Healthy Subject Studies to Assess the Effect of Different Electroacupuncture Parameters on Analgesia, Peripheral Sensory Thresholds and Central Pain Processing.
Brief Title: To Study the Mechanisms of Acupuncture Through Functional Magnetic Resonance Imaging and Peripheral Neurosensory Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: K08AT001695-01 (NIH); 050557
Record Dates: First submitted 2007-08-24; First posted 2007-08-28 (Estimated); Last update posted 2007-08-28 (Estimated); Status verified 2007-08

CONDITIONS: Healthy
Keywords: Acupuncture; Analgesia; Functional magnetic resonance imaging (fMRI); Neuronal Mechanisms; Quantitative Peripheral Sensory Testings; Normal Volunteers
MeSH Terms: conditions — Agnosia | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Electroacupuncture

SUMMARY:
Acupuncture may affect nerve functions. This study assesses the effect of acupuncture on both the peripheral and the central nerve systems

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80
* Male and female
* No acupuncture treatment for the past 2 weeks
* No analgesics for the past 2 weeks
* Absence of neuropathic pain states

Exclusion Criteria:

* History of psychological illness
* History of Claustrophobia
* Lack of ability to understand the experimental protocol and to adequately communicate in English
* Pregnancy
* Pending litigation
* History of head trauma
* History of trauma or surgery to lower extremities and pelvic area

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2003-09; Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Leung, M.D., Principal Investigator — University of California, San Diego
Locations (1):
- The University of California, San Diego, Medical Center, La Jolla, California, United States